CLINICAL TRIAL: NCT00442377
Title: Exposure of Human Volunteers to Live Malaria Sporozoites Under Chloroquine Prophylaxis
Brief Title: Study to Investigate the Induction of an Protective Immune Response to Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EHMI-8
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: Falciparum Malaria
Keywords: Falciparum; Plasmodium; Malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria

INTERVENTIONS:
Procedure: exposure to malaria sporozoites

SUMMARY:
The objective of the study is to induce a protective immune response against malaria in healthy human volunteers. The different parts of the immune response will then be studied.

DETAILED DESCRIPTION:
Efforts to develop vaccines against malaria still represent a substantial focus of current research activities. Factors that have hampered the development of a subunit vaccine include the complexity of the malaria life cycle, the wide variety of immune response induced by the malaria parasite, and an incomplete knowledge of protective immunity. This study is therefore aimed at inducing protective immunity against malaria in 15 healthy volunteers. Volunteers will be exposed to the bites of infectious mosquitoes 3 times with live P. falciparum sporozoites under chloroquine prophylaxis. Challenge with infected mosquitoes will be given after stopping chloroquine prophylaxis.

Five volunteers will form a control group; they will be exposed to non-infectious mosquitoes under chloroquine prophylaxis.

Endpoints include the time and height of parasitemia after challenge, the development of fever and immunological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 45 years healthy volunteers (males or females).
* General good health based on history and clinical examination.
* All volunteers have to sign the informed consent form.
* Negative pregnancy test.
* Use of adequate contraception for females
* Reachable by phone during the whole study period.
* Volunteer agrees to inform the general practitioner and agrees to sign a request for medical information concerning contra-indications for participation in the trial

Exclusion Criteria:

* History of malaria or residence in malaria endemic areas within the past six months.
* Positive serology for P. falciparum
* Previously participated in any malaria vaccine study
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers.
* Cardiovascular risk >10% according to European guidelines, taking into account sex, age, cholesterol, weight, smoking habits, blood pressure, diabetes
* Any laboratory abnormalities on screened blood samples beyond the normal range, as defined at UMC St Radboud. Positive HIV, HBV or HCV tests.
* Volunteers should not be enrolled in any other clinical trial during the whole trial period.
* Volunteers should not receive chronic medication, especially immunosuppressive agents (steroids, immunomodulating or immunosuppressive drugs) during the three months preceding the screening visit or during the study period.
* Pregnant or lactating women.
* Volunteers unable to give written informed consent.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study.
* Known hypersensitivity for anti-malaria drugs
* Volunteers are not allowed to travel to malaria endemic countries during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
A significant difference in time of thick smear positivity between exposed and control groups
A significant difference in parasitemia as measured by 18S Pf NASBA between exposed and control group
A significant difference in kinetics of parasitemia between exposed and control groups as measured by 18S Pf NASBA.
A difference in occurrence or height of fever between exposed and control groups.

SECONDARY OUTCOMES:
Significant differences in immune response between exposed and control volunteers (including NK-cell reactivity, TLR reactivity and regulatory T-cell reactivity)
Significant differences in the outcome of in vitro functional malaria assays between exposed and control volunteers
Significant differences in cellular reactivity against Pf antigens
Significant differences in parasite VAR gene expression during infection
The identification of immune mechanisms that correlate with protection
6. The identification of potential vaccine candidates that correlate with protection

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, Prof, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Coffeng LE, Hermsen CC, Sauerwein RW, de Vlas SJ. The Power of Malaria Vaccine Trials Using Controlled Human Malaria Infection. PLoS Comput Biol. 2017 Jan 12;13(1):e1005255. doi: 10.1371/journal.pcbi.1005255. eCollection 2017 Jan. PMID 28081133
- [Derived] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203